CLINICAL TRIAL: NCT02108626
Title: A Behavioral Assessment of Electronic Cigarettes in Reducing Cue- and Withdrawal-induced Craving in Daily Dependent Smokers
Brief Title: Electronic Cigarettes in Daily Dependent Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Laurie Zawertailo, Independent Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 001/2014
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Substance Withdrawal Syndrome; Nicotine Dependence
Keywords: Electronic Cigarettes; Lozenge; Nicotine; Tobacco; Dependence; Withdrawal
MeSH Terms: conditions — Substance Withdrawal Syndrome; Tobacco Use Disorder; Vaping | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- E-Cigarette with nicotine (Active Comparator): Electronic cigarette with cartridge fluid containing nicotine
  Interventions: Drug: Nicotine
- E-Cigarette without nicotine (Placebo Comparator): Electronic cigarette with cartridge fluid containing no nicotine (placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotine — E-Cigarette with nicotine cartridge
  Arms: E-Cigarette with nicotine
Drug: Placebo — E-Cigarette with 0mg nicotine cartridge
  Arms: E-Cigarette without nicotine

SUMMARY:
The aim of this study is to measure nicotine cue- and withdrawal-induced craving in current smokers under four distinct conditions: after smoking a conventional cigarette, an electronic cigarette (e-Cigarette) containing nicotine, an e-Cigarette without nicotine, and after taking a nicotine lozenge. Participants will be asked to attend four morning study visits after overnight smoking abstinence. Standardized questionnaires will be used to assess changes under each condition, allowing for the investigation of the efficacy of e-Cigarettes in reducing craving by replacing the behavioral component of smoking with minimal risk of adverse effects.

DETAILED DESCRIPTION:
Many addiction models postulate stimuli to be linked with nicotine intake and reward after prolonged use. As such, smoking becomes more heavily based in habit, initiated by cues. Craving has been found to be a crucial component of continued smoking and relapse in response to various environmental and behavioral cues. Electronic Cigarettes (e-Cigarettes) are new smoking products emerging in consumer markets that often mimic conventional tobacco cigarettes. E-Cigarettes commonly include a cartridge, a heating element, a puff sensor, and a battery. When a user draws on the device, the heating element is activated and the cartridge fluid is vaporized. Users then inhale the aerosol containing droplets of the vaporized fluid. This study will empirically assess the efficacy of e-Cigarettes in alleviating craving by replacing the behavioral component of smoking. Using standardized questionnaires, intra-subject changes in cue- and withdrawal-induced craving after smoking an e-Cigarette without nicotine will be compared with that after either smoking a conventional cigarette, an e-Cigarette with nicotine, or taking a 4mg lozenge.

ELIGIBILITY:
Inclusion Criteria:

* Current daily smoker
* Smoke minimum of 10 cigarettes per day
* Fagerstrom Test of Nicotine Dependence Score equal or greater than 3
* Never used an e-Cigarette prior to the study
* No intention to quit smoking within the next 3 months
* Able to provide written informed consent
* Able and willing to attend scheduled appointments

Exclusion Criteria:

* Any serious medical or unstable psychiatric problems requiring treatment
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Cue-induced nicotine craving | 1 hour after condition
  Craving assessment after presentation of smoking- and neutral-cues 1 hour after condition

SECONDARY OUTCOMES:
Withdrawal-induced nicotine craving | 3 hours after condition
  Craving assessment after presentation of smoking- and neutral-cues 3 hours after condition

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Zawertailo, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, BACDRL Lab, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Ng G, Attwells S, Selby P, Zawertailo L. Effectiveness of Non-Nicotinic E-Cigarettes to Reduce Cue- and Abstinence-Induced Cigarette Craving in Non-Treatment Seeking Daily Dependent Smokers. Psychopharmacology (Berl). 2021 Jun;238(6):1461-1472. doi: 10.1007/s00213-021-05772-4. Epub 2021 Jan 30. PMID 33515267
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre — http://www.camh.net/research